CLINICAL TRIAL: NCT02046018
Title: Healthy Child Uganda: Can Village Health Volunteers Trained in Integrated Community Case Management of Childhood Illness Improve Access to Care for Africa's Most Vulnerable Children?
Brief Title: Integrated Community Case Management (ICCM) Delivered by Village Health Teams in Bushenyi District in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Healthy Child Uganda (Other)
Responsible Party: Principal Investigator, Dr. Jenn Brenner, Clinical Associate Professor, Healthy Child Uganda
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HCU_AHSI
Record Dates: First submitted 2014-01-21; First posted 2014-01-27 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Maternal and Child Health
Keywords: Maternal and Child Health; Rural Uganda

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ICCM delivered by VHT (Active Comparator): Health Outcomes in Communities where VHT's were trained in ICCM and given drugs.
  Interventions: Other: ICCM delivered by VHT
- ICCM delivered by VHT with cell phone (Active Comparator): Health Outcomes in communities with VHT's who were trained in ICCM and given cell phones
  Interventions: Other: ICCM delivered by VHT; Other: ICCM delivered by VHT with Cell Phone
- Health outcomes in communities with no ICCM (Active Comparator): Health outcomes in communities with VHT's who were not trained in ICCM
  Interventions: Other: No intervention

INTERVENTIONS:
Other: ICCM delivered by VHT — VHT's deliver ICCM to children under five in their communities
  Arms: ICCM delivered by VHT; ICCM delivered by VHT with cell phone
Other: ICCM delivered by VHT with Cell Phone — ICCM delivered to children under 5 by VHT trained in ICCM and given cell phones
  Arms: ICCM delivered by VHT with cell phone
Other: No intervention — VHT's selected by no ICCM training given and no drugs or cell phones.
  Arms: Health outcomes in communities with no ICCM

SUMMARY:
In Sub-Saharan Africa (SSA), many children die from diarrhoea, acute respiratory illness (ARI) and malaria, despite well- recognized, inexpensive and highly effective treatments, since health access and human resources are limited. Healthy Child Uganda (HCU) is a Ugandan-Canadian partnership that since 2003, has developed, implemented and evaluated a Village Health Volunteer (VHV) program in 175 rural villages. Volunteers, selected by peers, provide health education and refer sick children. Volunteer retention (94%) and significant decreases in child deaths are remarkable. Now, HCU wonders whether VHV scope can extend to provide treatment for sick children using Oral Rehydration Salts (ORS)/Zinc, antibiotics, and antimalarials. Use of lay providers in this capacity, called integrated community case management (iCCM), has been proposed as a potential inexpensive solution to SSA's human health resource crisis.

PRIMARY QUESTION: In rural southwest Uganda, can iCCM provided by lay volunteers, improve the proportion of children with diarrhoea receiving ORS/Zn, ARI receiving antibiotics, and fever/malaria receiving antimalarials? Secondary study questions consider VHV capacity to prescribe appropriate drug, dose, duration; iCCM acceptance by family, and VHV; VHV retention/motivation; program cost. Selected VHV will be iCCM trained then receive treatments for distribution. Qualitative and quantitative methods including household surveys, and focus groups will consider pre/post intervention differences and differences in control and intervention populations. A research short course and micro research grants (~ $3000 to multidisciplinary groups pursuing relevant questions) will promote health system evaluation capacity. Lessons learned are critical as SSA countries move forward in planning for increased iCCM programming.

ELIGIBILITY:
Inclusion Criteria:

* Children under five (< or =59 months)

Exclusion Criteria:

* Children over five years (> 59 Months)

Max Age: 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5000 (Actual)
Dates: Start 2009-10; Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Percentage of change in number of children under five in intervention area who receive appropriate Integrated Community Case Management Treatment from a Community Health Worker for presumed pneumonia. | March 2013 - November 2014 (8 months)
  Children diagnosed by a Community Health Worker with presumed pneumonia (fast breathing and cough) treated with Amoxicillin.
Percentage of change in number of children under five in intervention area who receive appropriate Integrated Community Case Management Treatment from a Community Health Worker for diarrhea | March 2013 - November 2014 (8 months)
  Children diagnosed with diarrhea will be treated with ORS and zinc.
Percentage of change in number of children under five in intervention area who receive Integrated Community Case Management Treatment from a Community Health Worker for fever. | March 2013 - November 2014 (8 months)
  Children diagnosed with fever are presumed to have malaria, as per government treatment guidelines, and are treated with Coartem.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Maling, Principal Investigator — MUST; Celestine Barigye, Principal Investigator — MUST; Jerome Kabakyenga, Principal Investigator — MUST

REFERENCES:
- [Derived] Oliphant NP, Manda S, Daniels K, Odendaal WA, Besada D, Kinney M, White Johansson E, Doherty T. Integrated community case management of childhood illness in low- and middle-income countries. Cochrane Database Syst Rev. 2021 Feb 10;2(2):CD012882. doi: 10.1002/14651858.CD012882.pub2. PMID 33565123